CLINICAL TRIAL: NCT04156243
Title: Phase I, Interventional, Single Arm, Open Label, Treatment Study to Evaluate the Safety and Tolerability of CD19 CARvac in Patients With Relapsed and/or Refractory B Cell Malignancies
Brief Title: CD19 CARvac T Cells for Patients With Relapsed / Refractory B Cell Malignancies
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: iCell Gene Therapeutics (Industry)
Collaborators: Peking University Shenzhen Hospital (Other); Chengdu Military General Hospital (Other); iCAR Bio Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICG134-001
Record Dates: First submitted 2019-11-06; First posted 2019-11-07 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-01

CONDITIONS: B Cell Lymphoma; B Cell Leukemia
Keywords: CD19; CD19 CAR T cell
MeSH Terms: conditions — Lymphoma, B-Cell; Leukemia, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19 CARvac T cells (Experimental): CD19 CARvac T cells transduced with a lentiviral vector to express
  Interventions: Biological: CD19 CARvac T cells

INTERVENTIONS:
Biological: CD19 CARvac T cells — CD19 CARvac T cells administered to patients, will be either fresh or thawed CAR T cells by IV injection after receiving lymphodepleting chemotherapy.

SUMMARY:
This is a phase I, interventional, single arm, open label, treatment study to evaluate the safety and tolerability of CD19 CARvac in patients with relapsed and/or refractory B cell malignancies.

DETAILED DESCRIPTION:
CD19 CARvac is a chimeric antigen receptor immunotherapy treatment designed to treat

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis based on the World Health Organization (WHO) 2008
2. Patients have exhausted standard therapeutic options
3. Systematic usage of immunosuppressive drug or corticosteroid must have been stopped for more than 4 weeks
4. Female must be not pregnant during the study

Exclusion Criteria:

1. Prior solid organ transplantation
2. Potentially curative therapy including chemotherapy or hematopoietic cell transplant
3. Prior treatment with BCMAxCD3 or CS1xCD3 bispecific agents

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicity (DLT) as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | 28 days
Type of dose-limiting toxicity (DLT) | 28 days
Number of participants with adverse event by severity as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | 2 years

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 1 year
  Assessment of morphologic complete remission (CR), complete remission with incomplete recovery of counts (CR1), no residual disease as analyzed by flow cytometry analysis, and molecular remission by molecular studies
Progression-free survival (PFS) | 1 year
Overall survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hongyu Zhang, MD, PhD, Principal Investigator — Peking University Shenzhen Hospital; Fang Liu, MD, PhD, Principal Investigator — The General Hospital of Western Theater Command
Locations (2):
- China (2):
  - The General Hospital of Western Theater Command, Chengdu
  - Peking University Shenzhen Hospital, Shenzhen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu F, Sha S, Ma G, Su Y, Xiong Y, He G, Li Y, Hanes WM, Tse W. Treatment of CML-transformed B Cell Acute Lymphoblastic Leukemia (B-ALL) in Adults with Anti-CD19 Chimeric Antigen Receptor T Cell (CAR T) Therapy. Stem Cell Rev Rep. 2020 Dec;16(6):1356-1358. doi: 10.1007/s12015-020-10008-7. No abstract available. PMID 32840736